CLINICAL TRIAL: NCT02486783
Title: Infection, Sepsis and Meningitis in Surinamese Neonates
Acronym: InSepSur
Status: Completed | Type: Observational
Sponsor: Academic Hospital Paramaribo (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Rens Zonneveld, MD, Academic Hospital Paramaribo
Other Study IDs: VG 021-14A
Record Dates: First submitted 2015-06-27; First posted 2015-07-01 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Neonatal Sepsis; Neonatal Infection; Neonatal Meningitis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Baseline controls (no signs of infection): Neonates admitted for serial blood draws for uncomplicated hyperbilirubinemia
- Signs of infection A: No infection: antibiotics stopped after 48 hours; negative cultures
- Signs of infection B: Clinical infection: 7 day antibiotics; negative cultures
- Signs of infection C: Sepsis: positive bacterial blood culture
- Signs of infection D: Meningitis: positive bacterial CSF culture

SUMMARY:
Suriname is a small developing country in South America with a population of half a million people. Early neonatal death in Suriname is high with 16 per 1000 live births. Unpublished data from the Suriname Perinatal and Infant Mortality Survey estimate contribution of infection to early neonatal mortality at 25% (4 per 1000 live births) of all deaths. In comparison, incidence rates of neonatal sepsis alone are 3.5 per 1000 live births. These numbers indicate an increased burden of neonatal infection in Suriname versus the U.S. In any case about 40 newborns that die each year of infection are a huge loss, also considering the small Surinamese community. Despite this overall idea on the impact of infectious disease in Surinamese neonates exact information regarding incidence, type of infection (e.g., localized, viral, early-onset or late-onset sepsis), risk factors (e.g., insufficient antenatal care, maternal Group B-Streptococcus status), etiology, microbial causes, morbidity, antibiotic treatment (type and duration), and epidemiological determinants (e.g., gestational age, sex, ethnicity) are lacking.

From a clinical perspective, there is still a challenge to identify neonates with infection. Neonates are often admitted with ambivalent clinical symptoms and receive preventive antibiotics that are costly, promote pathogen-resistance, and have negative long-term effects (i.e., on the development of the intestinal bacterial flora). Currently, assessment of blood leukocyte or trombocyte counts and levels of CRP are insufficiently sensitive to be used as biomarkers, while confirmation of actual sepsis or meningitis by positive culture results is relatively rare (0.5-3% in the United States). This complicates decisions on duration of antibiotic treatment and hospitalization significantly, while no other biomarkers exist.

The circulating isoforms of adhesion molecules (cAMs), which mediate interactions of leukocytes with the vascular endothelium, have been proposed as biomarkers for infection and sepsis. During infection they accumulate in the bloodstream as a result of shedding, which represents their removal from cell surfaces of endothelial cells and leukocytes by enzymes called sheddases. Recently, we have reviewed mechanisms behind shedding of cAMs in neonatal, pediatric and adult sepsis. The shedding process reflects a critical and active process in orchestrating interaction between leukocytes and the endothelium for an effective host response, while minimizing collateral tissue damage. As a result, both plasma levels of cAMs and their sheddases are subject to change during infection and sepsis. Additionally, compelling, albeit limited, data suggest changes of levels of cAMs in CSF in adult and pediatric meningitis.

To date, some evidence exists of changes in levels of cAMs during malaria (in children from Malawi) and sepsis, although not sensitive enough to predict outcomes in the clinic. Those levels have never been assessed simultaneously with levels of their sheddases in blood or CSF as a diagnostic tool. We propose that this combined approach may provide more detailed information about the extent of inflammatory activation in neonates.While a balance in levels is maintained under resting conditions or mild (local) infection, it may be perturbed during sepsis or meningitis . Thus, simultaneous measurement of these levels could promote early identification of infection, and may even distinguish between mild infection, systemic infection or meningitis. Currently, manufacturers are rapidly developing Luminex® technology as an advanced, fast, high-throughput and clinically feasible bedside tool for such an approach.

We hypothesize that incidence rates of neonates with infection in Suriname are high. We further hypothesize that, upon signs of infection, the simultaneous measurement of cAMs and their SEs in serum and CSF discriminates between infected and non-infected neonates. We aim to: 1) identify and follow neonates at the Academic Hospital Paramaribo with signs of infection to establish incidence rates of infection, and 2) investigate diagnostic potential of our proposed biomarker combination in these neonates for infection, type of infection (e.g., local (mild), sepsis or meningitis) and outcomes.

DETAILED DESCRIPTION:
Study Design:

The Academic Hospital Paramaribo (AZP) has the largest perinatal care facility in Suriname. Recently, the AZP opened the country's only neonatal intensive care unit (NICU). This study aims to include all neonates presenting here and at the high and medium care facilities with clinical signs of infection, sepsis or meningitis (age: 0-1 month) that require infection work up. Along with the inclusion of these neonates follows a detailed epidemiological description of newborns with infectious disease. Inclusion will take place by one of 10 residents, with approval from one of the 5 attending pediatricians. Along with standard blood draws for infection parameters (at t=0 and t=48 hours), blood culture (at t=0 hours) and CSF culture (at t=0 hours), serum and CSF will be separated for our biomarker study. For all neonates, normal local protocol for the management of infection, sepsis or meningitis will be followed. This includes antibiotic treatment for 7 days when 1) clinical suspicion of infection at admission was high; 2) infection parameters are aberrant at 48 hours; 3) blood culture is positive. Otherwise, antibiotic treatment is stopped after 48 hours. Further protocol includes necessary changes in respiratory support, circulatory (fluid) support and feeding. Medical treatments can be cardiotonics and treatments for hyperglycemia and seizures. Neonates are divided over 5 groups based on course of antibiotic treatment and culture results: 1) Baseline controls (no signs of infection): neonates admitted for serial blood draws at t=0 and 48 hours for uncomplicated hyperbilirubinemia (with jaundice, but without other signs of infection); 2) Signs of infection, further divided in: 2a) No infection: antibiotics stopped after 48 hours; negative cultures; 2b) Clinical infection: 7 day antibiotics; negative cultures; 2c) Sepsis: positive bacterial blood culture; 2d) Meningitis: positive bacterial CSF culture.

Sample size and power:

Sample size and power analysis is complicated because The Suriname Perinatal and Infant Mortality Survey only provides data on mortality as a result of infection (amongst other causes), without data on the incidence of neonatal infection. We estimate an incidence of admission for clinical signs for infection of 50 per 1000 live births (5%) at the NICU of the AZP. An annual birth rate at the AZP of about 3000 live births per year gives us n=150 neonates with signs of infection divided over four groups. Based on these estimations the recommended sample size of the whole population would be n=1538 (margin of error 1% and CI 99%). Since the incidence of newborns for which exclusion criteria apply and incidence of the subgroups are currently unknown, and to compensate for loss to follow up, we decided to include over a one-year period (n=3000). The biomarker study is exploratory in nature and we aim for a baseline control group of n=40 (larger n may be difficult to establish due to practical constraint). In our analysis we will adjust for gestational age and ethnicity. Absence of prior data on levels of biomarkers in relation to neonatal infection prevents us from estimating power. With analysis of sera and CSF from our 150 inclusions we aim to perform that for future follow-up biomarker studies.

Methodology:

Epidemiology: The following data will be recorded upon (t=0 hours) and during (t=48 hours) admission: date and time, maternal age, gender, maternal Group-B-streptococcus culture result, maternal fever, (premature) prolonged rupture of membranes ((P)PROM), gestational age (if unknown according to Ballard), delivery location and mode, Apgar scores, birth weight, gender, ethnicity, leukocyte count and differentiation, trombocyte count, CRP, antibiotic treatment (type, duration), sepsis (early/late onset, line), survival/expiration. The Score for Neonatal Acute Physiology II will be scored at t=0 and 48 hours. .

Serum separation: Whole blood will be collected by vena puncture in one serum microtainer (500 μL). Serum samples will be separated by centrifugation at 2500 xg for 15 minutes and kept on ice until storage. All serum and CSF samples will be stored at -80°C in the central laboratory of the AZP. Batched serum and CSF samples will be packaged on dry-ice (max. 24 hours; according to the International Air Transport Association guidelines) and transported to the Endothelial Biomedicine and Vascular Drug Targeting Laboratory in Groningen.

Luminex® Technology: Our laboratory in Groningen has extensive experience with the use of Luminex® arrays for the measurement of multiple adhesion molecules at once in clinical patient samples (i.e., multiplexing). Currently, the technique is applied successfully in basic and translational research and is gradually making its way into the clinic, allowing for the compilation of a diagnostic multi-array of molecules for complex diseases, such as sepsis or cancer. See Table 1 for specific adhesion molecules and their associated shedding enzymes that we include in our array. Measurement of soluble L-, E-, and P-selectin, Intercellular adhesion molecule (ICAM-1), vascular cell adhesion molecule (VCAM-1), neutrophil elastase (NE), Matrix-metalloproteinase-9 (MMP-9), tissue-inhibitor of metalloproteinase (TIMP-1) and ADAM metallopeptidase domain 17 (ADAM-17) will be performed with Luminex®; NE and ADAM-17 will be analyzed by ELISA as long as Luminex® is not yet available for these molecules. We will also use Luminex® to measure circulating Angiopoetin-1 and -2, and soluble Tie-2 receptor as markers of endothelial cell activation. For Luminex® assays (Life Technologies) appropriate diluted volumes of samples will be aliquoted in 96 well plates. Simultaneous analysis will take place with the Luminex® 100 Analyzer (Life Technologies). ELISA will be performed according to the manufacturers protocol (R&D systems).

Statistical Analysis:

Incidence rates end epidemiological determinants will be calculated at the end of the inclusion period. Categorical variables will be presented as numbers and percentages and continuous variables as mean +/- SD or, if not normally distributed, as median +/- 10th percentile. Categorical data will be compared with chi-square and continuous variables with the independent t-test or two-way ANOVA. To assess the independent effect of biomarker combinations (cAM/SE ratios) on the occurrence of infections multivariate logistic regression will be performed with infection as dependent and cAM/SE ratios, gestational age and ethnicity as independent variables. We will calculate Spearman rank correlation to assess bivariable association between biomarkers. Diagnostic accuracy of cAM/SE ratios will be assessed by using the Receiver Operating Characteristic (ROC)-based area under the curve. Other test characteristics such as predictive value and likelihood ratios will be calculated. P-values < 0.05 will be considered statistically significant. Statistical analysis will be performed using Stata (StataCorp).

Difficulties and Limitations:

First, separation of serum from neonates could lead to low volumes, yet Luminex® technology is designed for the assessment of high numbers of molecules in low volumes. According to local protocol, CSF collection is not performed in baseline controls and not in neonates that are not suspect for meningitis. Measurement of two time-points may be insufficient to detect changes in time. We will not be able to identify viral causes of infection, since proper diagnostics are currently not available in Suriname.

Ethical concerns for the Surinamese situation:

We have received approval from the Surinamese Ethical Board on March 9th 2015. Upon eligibility of a newborn, at least one parent or guardian will be asked for participation of their child into the study and will be given written information in Dutch. If the patient is illegible or does not understand Dutch, oral explanation will be given in a language that is understood (either English or Sranan Tongo). Written informed consent (with either signature or fingerprint) is obtained from a parent or guardian for the collection of all clinical data, blood and CSF. Blood draws for serum separation and spinal tap for CSF collection will only take place along with interventions according to local protocol (i.e., no additional blood draws or spinal taps will take place). All samples will be treated anonymously and receive a sample ID.

Withdrawal of individual subjects:

Parents or guardians of subjects can initiate leave of the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject for medical reasons or when subjects are non-cooperative (i.e., resist blood draws).

Premature termination of the study:

There are no situations expected that would lead to premature termination of the study.

Safety reporting:

Adverse and serious adverse events population (base) We do not expect any (serious) adverse events related to drawing blood.

Administrative aspects and publication:

Handling and storage of data and documents: Paper data will be stored by the coordinating investigator, in a unique folder, which will be accessible by the coordinating investigator, and the investigators involved in the study. The data will also be stored electronically in an Excel database. The principal investigator will enter the data. The file will be only accessible by the investigators and data exchange through email will be encrypted with a password. Each participant will receive a unique participation number after signing informed consent, which corresponds to the sample ID of the blood sample.

Amendments:

Amendments are changes made to the research after a favorable opinion by the accredited ethical board has been given. All amendments will be notified that gave a favorable opinion. A 'substantial amendment' is defined as an amendment to the terms of the ethical board application, or to the protocol or any other supporting documentation, that is likely to affect to a significant degree:

* The safety or physical or mental integrity of the subjects of the trial;
* The scientific value of the trial;
* The conduct or management of the trial; or
* The quality or safety of any intervention used in the trial.

All substantial amendments will be notified to the ethical board and to the competent authority. Non-substantial amendments will not be notified to the accredited ethical board and the competent authority, but will be recorded and filed by the sponsor.

Annual progress report:

The sponsor/investigator will submit a summary of the progress of the study to the accredited ethical board once a year. Information will be provided on the date of inclusion of the first subject, numbers of subjects included and numbers of subjects that have completed the trial, serious adverse events/ serious adverse reactions, other problems, and amendments.

End of study report:

The investigator will notify the accredited ethical board of the end of the study within a period of 8 weeks. The end of the study is defined as the last patient's last visit. In case the study is ended prematurely, the investigator will notify the accredited ethical board, including the reasons for the premature termination. Within one year after the end of the study, the investigator/sponsor will submit a final study report with the results of the study, including any publications or abstracts of the study, to the accredited ethical board.

Public disclosure and publication policy:

The final publication of the study results will be written by the study coordinator(s) on the basis of the statistical analysis performed. A draft manuscript will be submitted to all co-authors for review. After revisions the manuscript will be sent to a peer reviewed scientific journal. The study coordinators must approve any publication, abstract or presentation based on patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

This study aims to include all neonates presenting here and at the high and medium care facilities with clinical signs of infection, sepsis or meningitis (age: 0-1 month) that require infection work up (i.e., laboratory testing and culturing):

* Baseline controls: uncomplicated jaunice, no other signs of infection
* Clinical signs of infection: tachypnea, dyspnea, apnea, grunting, tachycardia, bradycardia, hypotension, poor perfusion, vomitus, abdominal distension, constipation, poor feeding, lethargy, irritability, convulsions, temperature instability, pale, yellow, bleak, petechiae, bruising, bleeding.

Exclusion Criteria:

* Extreme prematurity: gestational below 32 weeks of gestational age
* Extreme dysmaturity: birthweight below 1500 grams
* Maternal HIV or malignancy

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns at the Academic Hospital Paramaribo without signs of infection (baseline controls) and with signs of infection admitted for infection work up and antibiotic treatment.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Presence of infection upon signs of infection | Within 7 days
  Descision on duration of antibiotics (48 hours or 7 days) and blood and liquor culture results

SECONDARY OUTCOMES:
Infection related mortality | 7 day and 30 day
Overall mortality due to infection | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Grietje Molema, PhD, Study Director — University Medical Center Groningen, The Netherlands
Locations (1):
- Academic Hospital Paramaribo, Paramaribo, Suriname

REFERENCES:
- [Background] Zonneveld R, Martinelli R, Shapiro NI, Kuijpers TW, Plotz FB, Carman CV. Soluble adhesion molecules as markers for sepsis and the potential pathophysiological discrepancy in neonates, children and adults. Crit Care. 2014 Feb 18;18(2):204. doi: 10.1186/cc13733. PMID 24602331
- [Derived] Zonneveld R, Jongman RM, Juliana A, Molema G, van Meurs M, Plotz FB. Serum concentrations of endothelial cell adhesion molecules and their shedding enzymes and early onset sepsis in newborns in Suriname. BMJ Paediatr Open. 2018 Oct 9;2(1):e000312. doi: 10.1136/bmjpo-2018-000312. eCollection 2018. PMID 30397669